CLINICAL TRIAL: NCT06145919
Title: Parent-Child Memory Study: Improving Future Thinking Among Mothers From a Traditionally Underserved Community to Reduce Harsh Parenting and Improve Child Outcomes - A Randomized Controlled Trial
Brief Title: Parent-Child Memory Study: Improving Future Thinking Among Mothers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: University of Kansas (Other); University of Maryland, College Park (Other); Michigan State University (Other)
Responsible Party: Principal Investigator, Melissa Maye, Principal Investigator; Associate Scientist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NHRCT: 16828-01
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Behavior, Health
Keywords: episodic future thinking; episodic recent thinking; delay discounting; parent-child relations; low resource; Flint, Michigan; special play time
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Episodic Future Thinking (EFT) (Experimental): Mothers will receive episodic future thinking (EFT). Mothers will meet with a "peer mother" who will administer the EFT intervention, including generation of several specific future events reflecting positive interactions with their child. The participant will be asked to discuss their relationship with their child and to give examples of both positive and negative parenting from their personal experience. The "peer mother" will then ask the participant to think about their long-term parenting goals and will discuss how to create a vivid event that will be easy to remember. We will also teach each parent a behavioral parent training element called Special Play Time. Following this session, participants are asked to engage in messaging that will prompt them to think about future events.
  Interventions: Behavioral: Episodic Future Thinking (EFT)
- Episodic Recent Thinking (ERT) (Active Comparator): In the episodic recent thinking (ERT) condition, the participant will be asked to discuss their relationship with their child and to give examples of both positive and negative parenting from their personal experience. The "peer mother" will then ask the participant to think about the present and discuss how to focus on the present. Two positive recent events and two negative recent events will be used to create ERT scenes for the parent to envision their current relationship with their child. We will also teach each parent a behavioral parent training element called Special Play Time. Following this session, participants will receive messages over the course of two weeks helping parents to focus on recent events with their child.
  Interventions: Behavioral: Episodic Recent Thinking (ERT)

INTERVENTIONS:
Behavioral: Episodic Future Thinking (EFT) — The adapted episodic future thinking (EFT) intervention will focus on generation of vivid, substance-free, rewarding events that could happen in the future with their children.
  Arms: Episodic Future Thinking (EFT)
Behavioral: Episodic Recent Thinking (ERT) — In the episodic recent thinking (ERT) condition, the participant will instead describe in vivid details events that have occurred in the recent past.
  Arms: Episodic Recent Thinking (ERT)

SUMMARY:
Parents of children from impoverished communities are disproportionately more likely to engage in harsh physical discipline, which can lead to serious clinical outcomes, including suicidal ideation and attempts. One mechanism linking low resource environments and maladaptive parenting strategies is maternal delay discounting, or the tendency to value smaller, immediate rewards (such as stopping children's misbehavior via physical means) relative to larger, but delayed rewards (like improving the parent-child relationship). This study will examine the efficacy of implementing a low-cost, brief intervention targeting the reduction of maternal delay discounting to inform broader public health efforts aimed at improving adolescent mental health outcomes in traditionally underserved communities.

DETAILED DESCRIPTION:
Harsh parenting is associated with serious and costly mental health problems among youth, including substance use, mood disorders, and suicidal ideation and behaviors. Of concern, these parenting practices are most common among families from impoverished communities; however, many behaviorally-based parenting interventions do not take into account the unique mechanisms linking environmental disadvantage to parenting approaches. While the causes of harsh parenting are complex and varied, one such mechanism may be parents' tendencies to prioritize immediate rewards (such as stopping a child's misbehavior via physical punishment like spanking and hitting) relative to larger, but delayed rewards (including improved parent-child relationship quality), known as delay discounting.

The aims of the current study are to conduct a Stage 1 parent-child dyad randomized control trial (RCT) (n = 72) examining the effectiveness of a brief, episodic future thinking (EFT) intervention in a community setting serving low-income mothers and additional implementation data. Participants will be randomized to receive either Episodic Future Thinking (EFT) or Episodic Recent Thinking (ERT) intervention arms. This case series will examine the efficacy of episodic future thinking (EFT) compared to episodic recent thinking (ERT) to target reduction of parenting-related delay discounting. Outcomes will evaluate the effect of EFT on reducing maternal delay discounting and harsh parenting and improving child clinical outcomes.

ELIGIBILITY:
Parent Inclusion Criteria:

1. A mother and or grandmother from the Flint area with a child/grandchild between the ages of 5-10 who can provide legal consent for that child
2. Self-report that they have consistent contact with the child/grandchild
3. Willing to participate in the study
4. Able to participate in written assessments and an intervention conducted in English
5. Have a working cell phone that can receive and send text messages and be willing to receive/send text messages as part of the study
6. Have a phone or device that's able to use video conferencing software if interested in virtual participation

Parent Exclusion Criteria:

1. Self-disclosed active suicidality/homicidality
2. Self-disclosed current bipolar disorder, schizophrenia, or psychosis
3. Self-reported current and ongoing involvement with child protective services

Child Inclusion Criteria:

1. Children must be between the ages of 5-10 and have a mother/grandmother willing to provide consent for their participation
2. Willing to participate in parent-child observation sessions
3. Elementary proficiency in English
4. Willing to participate in study surveys

Child Exclusion criteria:

1. Self-disclosed active suicidality/homicidality
2. Self-disclosed current bipolar disorder, schizophrenia, or psychosis

Min Age: 5 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 144 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Monetary Choice Questionnaire | Baseline, Intervention, Week 2, Month 3, Month 6, Month 9
  The Monetary Choice Questionnaire (MCQ) is a 27-item binary-choice task, which asks participants to select between two hypothetical monetary amounts: a smaller reward available immediately (e.g. $49 today) or a larger reward available after a delay (e.g. $60 in 89 days). The measure is scored to derive a discounting rate k, with larger values reflecting more problematic rates of discounting. Because k distributions are typically skewed, post-hoc natural logarithmic transformations will be performed, which have been shown to approximate normal distributions. The MCQ has been shown to have strong psychometric properties among adults and correlates with real rewards, as well as real-world risk behaviors.
Change in Consideration of Future Consequences Scale Score | Baseline, Intervention, Week 2, Month 3, Month 6, Month 9
  The Consideration of Future Consequences Scale1 (CFCS-14) is a 14-item self-report questionnaire that assesses active consideration of longer-term implications of an individual's actions. Lower scores on the CFCS-14 are associated with a greater focus on immediate needs and have been found to be associated with less engagement in health behaviors1819 and greater substance use. The measure has been used extensively among adult samples and demonstrates strong reliability and validity. Research suggests modest but significant correlations with the MCQ. Change in CFCS-14 score is measured by comparing scores at the post-intervention assessment timepoints with baseline scores.

SECONDARY OUTCOMES:
Change in Alabama Parenting Questionnaire Score | Baseline, Intervention, Week 2, Month 3, Month 6, Month 9
  Parents will report on their parenting styles and behavior using the Alabama Parenting Questionnaire (APQ). The APQ consists of five subscales that yield two broadband "positive" and "negative" parenting factors. The measure is widely used and validated among parenting populations. 42 items are ranked on a scale of 1-5 and scores are computed for each subscale (with possible scores ranging from 3-15 for corporal punishment to 10-50 for longer subscales including parental monitoring and involvement). Higher scores reflect greater levels of each subscore domain.
Change in Emotion Regulation Checklist | Baseline, Intervention, Week 2, Month 3, Month 6, Month 9
  Parents will report on children's emotion regulation using the Emotion Regulation Checklist (ECR). The ECR includes 24 items that yield two subscales: (1) lability/negativity and (2) emotion regulation. The measure is widely used and validated for parent-report of older children and young adolescents.

CONTACTS AND LOCATIONS:
Locations (1):
- Mothers of Joy Institute for Parenting and Family Wellness, Inc, Flint, Michigan, United States

REFERENCES:
- [Background] Felton JW, Collado A, Cinader M, Lejuez CW, Chronis-Tuscano A, Yi R. Exposure to maternal depressive symptoms and growth in adolescent substance use: The mediating role of delay discounting. Dev Psychopathol. 2021 Oct;33(4):1279-1289. doi: 10.1017/S0954579420000486. PMID 32519638
- [Background] Dassen FC, Houben K, Jansen A. Time orientation and eating behavior: Unhealthy eaters consider immediate consequences, while healthy eaters focus on future health. Appetite. 2015 Aug;91:13-9. doi: 10.1016/j.appet.2015.03.020. Epub 2015 Mar 23. PMID 25814191
- [Background] Felton JW, Collado A, Ingram KM, Doran K, Yi R. Improvement of Working Memory is a Mechanism for Reductions in Delay Discounting Among Mid-Age Individuals in an Urban Medically Underserved Area. Ann Behav Med. 2019 Oct 7;53(11):988-998. doi: 10.1093/abm/kaz010. PMID 30955043
- [Background] Lin H, Epstein LH. Living in the moment: effects of time perspective and emotional valence of episodic thinking on delay discounting. Behav Neurosci. 2014 Feb;128(1):12-9. doi: 10.1037/a0035705. PMID 24512061
- [Background] Moreland, A.M., Felton, J.F., Hanson, R.F., Jackson, C., & Dumas, J.E. (2016). The relation between parenting stress and parenting locus of control: Mechanisms of change in parenting interventions. Journal of Child and Family Studies, 25, 2046-2054.
- [Background] Snider SE, DeHart WB, Epstein LH, Bickel WK. Does delay discounting predict maladaptive health and financial behaviors in smokers? Health Psychol. 2019 Jan;38(1):21-28. doi: 10.1037/hea0000695. Epub 2018 Nov 26. PMID 30474996
- [Background] Stein JS, Wilson AG, Koffarnus MN, Daniel TO, Epstein LH, Bickel WK. Unstuck in time: episodic future thinking reduces delay discounting and cigarette smoking. Psychopharmacology (Berl). 2016 Oct;233(21-22):3771-3778. doi: 10.1007/s00213-016-4410-y. Epub 2016 Aug 23. PMID 27553824